CLINICAL TRIAL: NCT03508583
Title: Validity and Reliability of Turkish Version of Turkish Version of The Measure of Processes of Care (MPOC 56-20- SP)
Brief Title: Turkish Version of The Measure of Processes of Care (MPOC)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Duygu Turker, Principal Investigator, Hacettepe University
Other Study IDs: 46418926
Record Dates: First submitted 2018-04-07; First posted 2018-04-26 (Actual); Last update posted 2018-04-27 (Actual); Status verified 2018-04

CONDITIONS: Cerebral Palsy; Muscular Dystrophies; Autism Spectrum Disorder; Traumatic Brain Injury; Down Syndrome; Disability, Developmental; Disability Physical
Keywords: mpoc; Validity and Reliability
MeSH Terms: conditions — Cerebral Palsy; Muscular Dystrophies; Autism Spectrum Disorder; Brain Injuries, Traumatic; Down Syndrome; Developmental Disabilities

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participation: Parents will complete the The Measure of Processes of Care 56- 20 (MPOC 56-20) questionary
  Service providers will complete The Measure of Processes of Care for Service Providers (MPOC-SP)
  Interventions: Other: Participation

INTERVENTIONS:
Other: Participation — The mpoc 56 and mpoc 20 will be field-tested with a sample of 300 parents of children with disabilities residing in the Turkey.
  Professionals working with children with disabilities will be assessed with MPOC SP questionnaires

SUMMARY:
Family-centred care (FCS) is considered the best practice in providing rehabilitation to children with disabilities and special needs. Family-centred care has been described as a partnership approach to healthcare decision making. As a philosophy of healthcare, today many multidisciplinary healthcare facilities have organized their services according to a family-centred approach. TheMeasure of Processes of Care (MPOC) is the most widely used instrument to assess parents' self-reported experiences of family-centred behaviours of rehabilitation services providers. The aim of this study is to translate the scale to Turkish and to determine validity and reliability of The Measure of Processes of Care (MPOC 56- 20- SP)

DETAILED DESCRIPTION:
The MPOC is a questionnaire designed to find out what parents of children with disabilities think of the services they and their children receive and how these services affect their psychosocial outcome. MPOC exists in two versions: the 56-item version was published in 1995 and the MPOC-20 in 2004. The20-item version was developed due to disadvantage of the longer version, because its completion can be very time consuming and the consequences of low respondent percentages . King and colleagues assert that the56-item MPOC is useful for research, while the MPOC-20 is better applied as a measure of parents' perceptions of the elements of FCS. The 20 items in the short version are distributed among the same ﬁve scales as in the MPOC-56. This ensures that the MPOC-56/20 captures aspects of care and services that have most importance for parents. The items are included in one of the following ﬁve scales:

1 Enabling and partnership; 2 Providing general information; 3 Providing speciﬁc information about the child; 4 Coordinated and comprehensive care; 5 Respectful and supportive care.

The Measure of Processes of Care for Service Providers (MPOC-SP) was developed to assess FCS from the perspective of professionals. The MPOC-SP has also been used in many different studies with different populations.

ELIGIBILITY:
Inclusion Criteria:

* To be diagnosed as disabilities and special needs
* Pediatric service providers who agree to participate to study

Exclusion Criteria:

* Children whose family didn't accept to participate to study

Ages: 5 Years to 25 Years | Sex: All
Age Groups: Child, Adult
Study Population: The subjects will be recruited from children who lives in Turkey and, attend special education centers and hospitals.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2018-06-01 (Estimated); Study Completion 2019-08-01 (Estimated)

PRIMARY OUTCOMES:
The Measure of Processes of Care (MPOC- 56) | MPOC 56 was administered twice within a period of 1 week to participants in order to test the test-retest reliability of the scale.
  Assessing of the participation level of children. The Measure of processes of care-56 (MPOC 56) will be applied for once for 300 participants. The MPOC consists of 56 questions, which are related to important aspects of care that are closely related with satisfaction of parents. The 56 items are divided into ﬁve factorially deﬁned subscales: Enabling and Partnership (EP), ProvidingGeneral Information (PGI), Providing Speciﬁc Informationabout the Child (PSI), Coordinated and Comprehensive Care(CCC) and Respectful and Supportive Care (RS). The items are answered on a seven-point scale ranging from 7 ('to a very greatextent') to 1 ('not at all'), with a 0 for 'Not applicable'. A higherscore reﬂects a more favourable judgement of the care process.
The Measure of Processes of Care 20 (MPOC- 20) | MPOC 20 was administered twice within a period of 1 week to participants in order to test the test-retest reliability of the scale.
  The measure of processes of care consists of 20 questions, which are related to important aspects of care that are closely related with satisfaction of parents. The 20 items are divided into ﬁve factorially deﬁned subscales: Enabling and Partnership (EP), ProvidingGeneral Information (PGI), Providing Speciﬁc Informationabout the Child (PSI), Coordinated and Comprehensive Care(CCC) and Respectful and Supportive Care (RS). The items are answered on a seven-point scale ranging from 7 ('to a very greatextent') to 1 ('not at all'), with a 0 for 'Not applicable'. A higherscore reﬂects a more favourable judgement of the care process.
The Measure of Processes of Care for services providers (MPOC- SP) | MPOC SP was administered twice within a period of 1 week to participants in order to test the test-retest reliability of the scale.
  Self-assessment tool for pediatric service providers that measures the extent to which the services they provide are family-centred. The Measure of Processes of Care for Service Providers consists of 27 items categorized into four scales: (1) Showing Interpersonal Sensitivity (SIS), (2) Providing General Information (PGI), (3) Communicating Specific Information about the Child (CSI), and (4) Treating People Respectfully (TPR), .All response options are labelled, ranging from 1 ('never') to 7 ('to a great extent'). A higherscore reﬂects a more favourable judgement of the care process.

SECONDARY OUTCOMES:
Child Health Questionnaire - Parent Form 50 | At baseline]
  Assessing health-related quality of life of children

CONTACTS AND LOCATIONS:
Overall Officials: Mintaze Kerem Günel, prof.dr, Study Chair — Hacettepe University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dyke P, Buttigieg P, Blackmore AM, Ghose A. Use of the measure of process of care for families (MPOC-56) and service providers (MPOC-SP) to evaluate family-centred services in a paediatric disability setting. Child Care Health Dev. 2006 Mar;32(2):167-76. doi: 10.1111/j.1365-2214.2006.00604.x. PMID 16441851
- [Background] Hagen AK, Bjorbaekmo WS. Parents evaluation of the processes of care in child rehabilitation: a reliability study of the Norwegian translation of MPOC-20. Child Care Health Dev. 2012 Jan;38(1):48-53. doi: 10.1111/j.1365-2214.2010.01192.x. Epub 2010 Dec 28. PMID 21198778
- [Background] Bjerre IM, Larsson M, Franzon AM, Nilsson MS, Stromberg G, Westbom LM. Measure of Processes of Care (MPOC) applied to measure parent's perception of the habilitation process in Sweden. Child Care Health Dev. 2004 Mar;30(2):123-30. doi: 10.1111/j.1365-2214.2003.00403.x. PMID 14961865